CLINICAL TRIAL: NCT00051376
Title: Vascular Interaction With Age in Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 154; R01HL070059 (NIH)
Record Dates: First submitted 2003-01-09; First posted 2003-01-13 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-11

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Arginine

INTERVENTIONS:
Drug: L-Arginine

SUMMARY:
The body produces a natural compound, nitric oxide (NO), which is known to improve the elasticity of blood vessels effect cardiac function and play a role in the remodeling process after a heart attack. The primary source of NO is one of the amino acids that the body uses to form new proteins, L-Arginine; although many individuals with heart disease also take medicines to increase the concentrations of NO such as nitroglycerine. The VINTAGE-MI trial is intended to investigate wether supplementation of the bodies supply of NO with oral administration of L-Arginine will improve the functional recovery of older patients who have recently suffered their first heart attack.

DETAILED DESCRIPTION:
BACKGROUND:

As we age, both our blood vessels and heart muscle naturally become stiff and loose their ability to flex as the heart beats and blood pressure changes. This is believed to worsen both blood vessel and cardiac function in older individuals. The stiffened tissue is likely to be less able to adapt to the stresses and remodeling that occur after a heart attack (myocardial infarction) because the loss of functional heart tissue predisposes the heart to poor function and the hearts blood vessels undergo various changes in order to increase the supply of blood to the damaged areas.

DESIGN NARRATIVE:

VINTAGE-MI is a randomized, double blind study enrolling patients who have recently suffered their first heart attack. There are two recruitment clinics within the Johns Hopkins University Network, the Johns Hopkins Hospital and the Hopkins Bayview Medical Center. Following preliminary testing to establish eligibility and baseline function of both the heart and blood vessels, study participants will be randomly assigned to receive either L-Arginine or a placebo pill which is identical except that it does not contain L-Arginine. These pills will be taken orally 3 times a day for 6 months. Participants will return to the clinic 1, 3, and 6 months after they begin taking their medication to have the same functional testing repeated.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Patients will have suffered their first acute Q-wave MI within 3 to 21 days with creatine kinase levels 3 times normal. All patients will have systolic blood pressure over 100 mmHg and the permission of their attending physician and the ability to give voluntary informed consent. Patients will be excluded if they have had a prior Q-wave infarction, present cardiogenic shock, unstable angina or non-cardiac disease limiting life expectancy to less than 1 year. Other exclusion criteria include significant kidney or liver disease, uncontrolled diabetes, or symptomatic cerebrovascular disease (such as stroke). Patients who have been previously shown to be non-compliant will be asked not to participate.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schulman — Johns Hopkins University

REFERENCES:
- [Result] Schulman SP, Becker LC, Kass DA, Champion HC, Terrin ML, Forman S, Ernst KV, Kelemen MD, Townsend SN, Capriotti A, Hare JM, Gerstenblith G. L-arginine therapy in acute myocardial infarction: the Vascular Interaction With Age in Myocardial Infarction (VINTAGE MI) randomized clinical trial. JAMA. 2006 Jan 4;295(1):58-64. doi: 10.1001/jama.295.1.58. PMID 16391217